CLINICAL TRIAL: NCT02256215
Title: Vitamin D in the Treatment of Primary Restless Legs Syndrome: 12 Weeks, Triple-blinded, Randomized, Placebo-controlled Trial
Brief Title: Vitamin D in the Treatment of Primary Restless Legs Syndrome
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Abdulaziz University (Other)
Collaborators: King AbdulAziz City for Science and Technology (Other)
Responsible Party: Principal Investigator, Siraj Omar Wali, Assistant professor, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RLSD-1234
Record Dates: First submitted 2014-10-01; First posted 2014-10-03 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Restless Legs Syndrome
Keywords: Vitamin D
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Vitamin D (Experimental): • All patients will have their serum vitamin D levels measured at the baseline visit. Those assigned to the treatment arm (group A) will receive either 50,000 international units of vitamin D3 by mouth once or more per week for six to eight weeks, then 800 to 1000 (or more) international units of vitamin D3 daily thereafter, this is according to the recommendations of the Endocrine Society clinical practice guideline 2011. Group B patients will receive placebo supplements identical in appearance to the vitamin D supplements.
  Interventions: Drug: Vitamin D
- Placebo (Placebo Comparator)

INTERVENTIONS:
Drug: Vitamin D
  Arms: Vitamin D

SUMMARY:
Restless Legs Syndrome (RLS) is a sensorimotor disorder that syndrome may substantially interfere with normal sleep, leading to significant impairment in patients' productivity and quality of life.

The most common and potent of all treatment regimens are the dopaminergic agonist agents, which carry serious adverse events in their prolonged use despite their augmentation. A few basic studies have suggested a potential relationship between vitamin D and RLS. It has been implicated that dopaminergic system dysfunction plays a role in the development of RLS, while vitamin D has a protective effect on that system. This has been further substantiated by few clinical observations that showed prompt improvement of RLS patients upon receiving dopaminergic agents such as carbamazepine. Other studies have revealed low serum levels of vitamin D in RLS patients, along with remarkable improvement after vitamin D replacement therapy, as has been demonstrated in a recent pilot study.

This collectively points at vitamin D as a potential, more natural and safer treatment option for those suffering from RLS. However, the role of vitamin D in RLS has not been effectively investigated. The aim of this 12-week, triple-blinded, randomized, placebo-controlled trial is to confirm the relationship between vitamin D deficiency and RLS and hence elucidate the efficacy of vitamin D replacement therapy in reducing the severity of RLS, with predictions that the results will contribute to better understanding of the disease and its management.

Methods and Materials: This 12-week, double-blinded, randomized, placebo-controlled trial is take place over a duration of 2 years. It will be held in the city of Jeddah to assess a sample of Saudi residents of the Western region.

It is comprised of a number of visits, with the first one consisting of a questionnaire that is to be answered regarding RLS, physical examination, electromyography, the objective multiple Suggested Immobilization test, and blood tests. The main purpose of the second visit is to establish a diagnosis of RLS.

Clinic visits number 3 through 6 comprise the pre-randomizaiton phase. Their purpose is to determine the patient's adherence to trial procedures and pharmacological treatment.

Then, patients are to visit the clinic every two weeks for the first two months, then at week 12. Patients will be assessed in regards to treatment response and adverse effects through history and physical examination along with further blood tests.

Aim: to confirm the relationship between vitamin D deficiency and RLS and hence elucidate the efficacy of vitamin D replacement therapy in reducing the severity of RLS, with predictions that the results will contribute to better understanding of the disease and its management.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed or already diagnosed patients with primary RLS and vitamin D deficiency.
2. Patients that are not currently receiving any treatment for RLS or vitamin D replacement therapy.
3. Patients from 18 to 75 years old.
4. Patients otherwise are in good general health.

Exclusion Criteria:

1. Patients diagnosed with secondary RLS. i.e.: patients with:

1. Iron deficiency anemia 2. End-stage renal disease. 3. Diabetes mellitus (DM). 4. Peripheral neuropathy. 5. Multiple sclerosis (MS). 6. Pregnancy.

2. Patients with other mimicking disorders or primary sleep disorders. E.g.:

1. Arthritis.
2. Deep venous thrombosis.
3. Varicose veins or venous insufficiency.
4. Habitual foot tapping.

3. Patients receiving medications that can trigger RLS. i.e.:

1. Anti hypertensive medications. E.g. Use of thiazide diuretics at a total dose greater than 37.5 mg/day.
2. Anti convulsion medications.e.g. Use of anticonvulsant drug started within 6 months of screening. Stable regimen of anticonvulsants is allowed.
3. Antinausea drugs (prochlorperazine or metoclopramide).
4. Antipsychotic drugs (haloperidol or phenothiazine derivatives).
5. Anti depressants (SSRIs).
6. Antihistamines as in cold and allergy medications.

4. Patients with current medications or conditions that would interfere with vitamin D absorption:

1. Celiac disease. 2. Chron's disease. 3. Chronic pancreatitis. 4. Cystic fibrosis. 5. Weight-loss drug e.g. orlistat. 6. Cholesterol-lowering drug e.g. cholestyramine

5. Patients with contraindications for vitamin D supplements. i.e.:

1. Hyperparathyroidism.
2. Kidney stones.
3. Liver diseases.
4. Granulomatous disorders (sarcoidosis, tuberculosis)

6. Patients 17 years old and younger.

7. Use of supplements containing vitamin D at total doses higher than 1000 IU/day within 12 weeks of the baseline visit initiating the protocol and unwillingness to limit vitamin D supplementation dosage to no higher than 1000 IU/day for the duration of the study.

8. Use of supplements containing calcium at total doses higher than 600 mg/day within 1 week of the baseline visit initiating the protocol and unwillingness to limit calcium supplementation dosage to no more than 600 mg/day for the duration of the study.

9. History of intolerance to vitamin D supplements.

10. Women only: A. Pregnancy (past 1 year by report or positive pregnancy test at screening), intent to become pregnant in the next 4 years or unprotected intercourse. History of gestational diabetes is not an exclusion criterion.

B. Currently breastfeeding. C. Use of oral contraceptives or menopausal hormone therapy started within 3 months of baseline. Stable regimen of oral contraceptives or any other hormonal method of contraception (e.g. implantable) is allowed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in The International Restless Legs Scale (IRLS) total score | 12 weeks

REFERENCES:
- [Derived] Wali SO, Abaalkhail B, Alhejaili F, Pandi-Perumal SR. Efficacy of vitamin D replacement therapy in restless legs syndrome: a randomized control trial. Sleep Breath. 2019 Jun;23(2):595-601. doi: 10.1007/s11325-018-1751-2. Epub 2018 Nov 14. PMID 30430372